CLINICAL TRIAL: NCT03816540
Title: Diaphragmatic Breathing and Heart Rate Variability Training for Improving Hypertension in Fragile X Associated Tremor/Ataxia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: UC Davis MIND Institute (Unknown); UC Davis, Mini-Grant Geriatrics (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1151848
Record Dates: First submitted 2018-05-08; First posted 2019-01-25 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Hypertension; FXTAS
MeSH Terms: conditions — Hypertension; Fragile X Tremor Ataxia Syndrome

STUDY DESIGN:
Intervention Model Description: Same intervention will be applied to FXTAS-affected and unaffected (comparison) participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FXTAS-affected (Experimental): FXTAS-affected participants will receive HRV and respiratory coherence biofeedback training for 20 sessions.
  Interventions: Device: HRV and respiratory coherence biofeedback
- FXTAS-unaffected (Active Comparator): FXTAS-unaffected participants will be assessed to compare the effects of biofeedback based on FXTAS status. This arm will receive HRV and respiratory coherence biofeedback training for 20 sessions.
  Interventions: Device: HRV and respiratory coherence biofeedback

INTERVENTIONS:
Device: HRV and respiratory coherence biofeedback — Biofeedback treatment to support self-regulatory processes on the physiological level: heart rate variability (HRV) and respiratory coherence.

SUMMARY:
To study whether heart rate variability training and respiratory coherence can improve hypertension in individuals with FXTAS.

All patients will receive HRV biofeedback training for 20 sessions. Our hypothesis is that individuals with FXTAS who undergo 20 sessions of biofeedback training will improve self-regulatory skills for reducing hypertension, as measured by blood pressure measurement to below 140/90. The investigators hypothesize that individuals who successfully develop increased heart rate variability and better synchrony between heart rhythm and respiration will show the greatest improvements in self-regulatory skills for hypertension.

DETAILED DESCRIPTION:
Fragile X-associated tremor ataxia syndrome (FXTAS) is a late onset neurodegenerative disease that affects carriers of the fragile X premutation. This project proposes the evaluation of an innovative intervention program that promotes self-regulatory skills for hypertension in individuals with FXTAS. Using a control-group experimental design, the investigators propose to explore the efficacy of a biofeedback treatment to support self-regulatory processes on the physiological level: Heart Rate Variability (HRV) and respiratory coherence biofeedback.

Chronic hypertension contributes to cardiovascular complications, dementia, and increased risk of stroke. Our results indicate that the risk of hypertension is significantly elevated in male premutation carriers with FXTAS compared with carriers without FXTAS and controls.

Several research studies showed high levels of physiological arousal in individuals with Fragile X-Associated Disorders (FXS/FX-AD), related to a dysregulation of the sympathetic and parasympathetic nervous system. One parameter to measure physiological arousal is cardiovascular activity. It provides an index of parasympathetic and sympathetic involvement of the autonomic nervous system. Heart rate is under the control of efferent sympathetic and vagal activities directed to the sinus node, which are modulated by central brain stem (vasomotor and respiratory centers) and peripheral oscillators (oscillation in arterial pressure and respiratory movements). Spectral analysis of heart rate variability (HRV) is a reliable quantitative method for analyzing the modulatory effects of neural mechanisms on the sinus node.

Biofeedback treatments are reported for over 30 years. Biofeedback provides specific information about internal biological processes (i.e. muscle activity, respiration, heart rate variability, skin temperature and brain electrical activity) in an individual. In general, by enhancing the awareness of these processes and training to volitional control over them, specific parameters can be improved. The internal biological processes can be measured with a specific biofeedback equipment that convert this data into signals, often in the form of auditory, visual or somatosensory events, so that the individual can perceive real-time changes in their physiological activity. As the individual learns to control these events, healthier physiological processes are conditioned. Depending upon the physiological processes targeted, healthier patterns of activity can be achieved by most people after they have participated in 10 to 50 sessions of biofeedback supported with professional coaching and practice. Various biofeedback protocols and assistive electronic technologies such as the NeXus-10, emWave Personal Stress Reliever® or StressEraser® exist to enhance the balance of parasympathetic activity, vagal tone, increase HRV and synchronize respiration with the heart rhythm (i.e., the slowing down and speeding up of the heart over time).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 50-90 with a molecular documentation of a fragile X premutation, diagnosed with FXTAS.
2. stable current pharmacological treatment regimen for at least 4 weeks.
3. English speaking (the intervention is currently only available in English)
4. Clinically significant hypertension.
5. Normal or corrected to normal vision and hearing.

Exclusion Criteria:

1. Significant medical and behavioral problems that would interfere with the study (e.g. not being able to sit and play a computer game for 10 minutes)
2. Participants who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study
3. Individual is non-verbal (has no spoken language)
4. English is not the primary language.
5. Clinically critical Hypertension that requires medical attention

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure (systolic & diastolic) | Baseline, 4 to 6 weeks
  Blood pressure is measured at the brachial artery of left arm using an electronic blood pressure monitor with an inflatable cuff, repeated three times at each site, and averaged. Less than 120/80 mmHg is considered "normal," 120/80 to 139/89 mmHg is "prehypertension," and above 140/90 mmHg is "hypertension."
Clinical Global Impression Scale - Severity (CGI-S) | Baseline
  The CGI-Severity (CGI-S) will be assessed at baseline according to the severity of hypertension, which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline elevated; 3=mildly elevated; 4=moderately elevated; 5=markedly elevated; 6=severely elevated; 7= extremely elevated. This rating is based upon observed and reported symptoms, behavior, and function in the past seven days. Symptoms and behavior can fluctuate over a week; the score should reflect the average severity level across the seven days.
Clinical Global Impression Scale - Improvement (CGI-I) | 4 to 6 weeks
  The CGI-Improvement (CGI-I) is similar to the CGI-S. Directly post-treatment and at the follow-up, the investigator compares the patient's overall clinical condition to the one week period just prior to the baseline visit. The query hypertension is rated on a seven-point scale: "Compared to the patient's condition at baseline, this participant's condition is: 1=very much improved since the baseline; 2=much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6= much worse; 7=very much worse since the baseline measure.

SECONDARY OUTCOMES:
Psychophysiological Profile - Heart Rate Variability (HRV) | 4 to 6 weeks
  HRV will be assessed using the emwave2 desktop device (HeartMath Institute, Boulder Creek, CA). It uses an earlobe plethysmograph sensor to detect the pulse wave, and plots changes in heart rate on a beat-to-beat basis.
Psychophysiological Profile - Synchrony between Respiration and HRV | 4 to 6 weeks
  A measure of synchrony will be assessed which will be calculated using the HRV measure previously described and respiration, which will be recorded by strain gauges placed around the abdomen.
Psychophysiological Profile - Skin Conductance | 4 to 6 weeks
  Galvanic skin response is measured in Siemens by the skin's conductance between two small metal electrodes placed on the walls of the index finger tip and the ring finger tip.
Mini-Mental State Examination (MMSE) | 4 to 6 weeks
  The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley RT, McCraty R, Atkinson M, Tomasino D, Daugherty A, Arguelles L. Emotion self-regulation, psychophysiological coherence, and test anxiety: results from an experiment using electrophysiological measures. Appl Psychophysiol Biofeedback. 2010 Dec;35(4):261-83. doi: 10.1007/s10484-010-9134-x. PMID 20559707
- [Background] Lehrer PM, Vaschillo E, Vaschillo B. Resonant frequency biofeedback training to increase cardiac variability: rationale and manual for training. Appl Psychophysiol Biofeedback. 2000 Sep;25(3):177-91. doi: 10.1023/a:1009554825745. PMID 10999236
- [Background] Lloyd A, Brett D, Wesnes K. Coherence training in children with attention-deficit hyperactivity disorder: cognitive functions and behavioral changes. Altern Ther Health Med. 2010 Jul-Aug;16(4):34-42. PMID 20653294
- [Background] Hamlin AA, Sukharev D, Campos L, Mu Y, Tassone F, Hessl D, Nguyen DV, Loesch D, Hagerman RJ. Hypertension in FMR1 premutation males with and without fragile X-associated tremor/ataxia syndrome (FXTAS). Am J Med Genet A. 2012 Jun;158A(6):1304-9. doi: 10.1002/ajmg.a.35323. Epub 2012 Apr 23. PMID 22528549
- [Background] Pagani M, Rimoldi O, Pizzinelli P, Furlan R, Crivellaro W, Liberati D, Cerutti S, Malliani A. Assessment of the neural control of the circulation during psychological stress. J Auton Nerv Syst. 1991 Jul;35(1):33-41. doi: 10.1016/0165-1838(91)90036-3. PMID 1940025
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Lubar JF, Bahler WW. Behavioral management of epileptic seizures following EEG biofeedback training of the sensorimotor rhythm. Biofeedback Self Regul. 1976 Mar;1(1):77-104. doi: 10.1007/BF00998692. PMID 825150